CLINICAL TRIAL: NCT02528617
Title: The Effect of Velaglucerase Alfa (Vpriv) on Skeletal Development in Pediatric Gaucher Disease
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No subjects accrued and no potential subjects were identified..
Sponsor: Baylor Research Institute (Other)
Collaborators: Texas Scottish Rite Hospital for Children (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 014-285
Record Dates: First submitted 2015-07-28; First posted 2015-08-19 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Gaucher Disease Type 1; Gaucher Disease Type 3
MeSH Terms: conditions — Gaucher Disease | interventions — Glucosylceramidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gaucher Type 1 or 3 (Other): Velaglucerase alfa IV 60 units/kg every other week for duration of the study.
  Interventions: Drug: Velaglucerase alfa

INTERVENTIONS:
Drug: Velaglucerase alfa — Enzyme replacement therapy
  Other Names: VPRIV

SUMMARY:
The purpose of this trial is to study the effect of Velaglucerase Alfa on skeletal bone development of children with Type 1 or Type 3 Gaucher Disease. In addition, the natural history and neurological status of children with Type 3 Gaucher Disease will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Enzyme Replacement Therapy naive,
* confirmed diagnosis of Gaucher disease type 1 or 3,
* able to travel to Dallas, Texas 1x per year for baseline plus 3 consecutive years,
* able to tolerate all study procedures,
* skeleton not fully formed as confirmed by DXA and MRI),
* and willing to receive velaglucerase alfa infusions every other week for the duration of the study.

Exclusion Criteria:

* Clinically unstable,
* taking or have taken bisphosphonates,
* Gaucher type 2,
* pregnant female,
* or deemed inappropriate for participation by the principal investigator.

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2015-07 (Estimated); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change in Z-scores from baseline in Skeletal Bone Mineral Density by Duel-energy X-ray absorptiometry (DXA) in children with Gaucher Disease type 1 and 3 receiving velaglucerase alfa. | Baseline pre-intervention and yearly thereafter for 3 years

SECONDARY OUTCOMES:
Change in degrees/second from baseline in saccadic eye movements in children with Gaucher type 3 receiving velaglucerase alfa. | Baseline pre intervention and yearly thereafter for 3 years
Change from baseline neurodevelopmental testing normalized scores in children with Gaucher Disease type 3 receiving velaglucerase alfa. | Baseline pre intervention and yearly thereafter for 3 years
Change from baseline brainstem auditory evoked potential results measured in microvolts in children with Gaucher Disease type 3 receiving velaglucerase alfa. | Baseline pre-intervention and yearly thereafter for 3 years
Change from baseline EEG (electroencephalogram) results measured in Hertz in children with Gaucher Disease type 3 receiving velaglucerase alfa. | Baseline pre-intervention and yearly thereafter for 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Schiffmann, M.D.,M.H.Sc., Principal Investigator — Baylor Research Institute/Institute of Metabolic Disease
Locations (1):
- Baylor Research Institute, Dallas, Texas, United States